CLINICAL TRIAL: NCT00946114
Title: A Local, Multi-Centre, Open Label Access Study, To Provide Sildenafil Therapy To Eligible Adult Patients With Pulmonary Arterial Hypertension For One Hundred Twelve Weeks / Prior To Reimbursement And Availability For Patients In Poland.
Brief Title: To Provide Sildenafil Therapy To Eligible Adult Patients With Pulmonary Arterial Hypertension For 112 Weeks
Status: Completed | Type: Observational
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A1481242
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Results first posted 2010-03-30 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: sildenafil — tablets, 20mg, TID, 112 weeks at the maximum
Drug: sildenafil — tablets, 20mg x 4 (80mg), TID, approximately 70 weeks

SUMMARY:
The purpose of this study is to provide sildenafil therapy to eligible adult patients with pulmonary arterial hypertension (PAH) and to the patients who completed the A1481142 study for the treatment of PAH in Poland. Only safety and tolerability data will be collected in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 and over who have any of the following conditions:

   * Idiopathic pulmonary arterial hypertension.
   * PAH associated with connective tissue disease (CTD).
   * PAH with surgical repair, at least 5yrs previously, of atrial septal defect (ASD), ventricular septal defect (VSD) patent ductus arteriosis (PDA) or aorta-pulmonary window.
2. Subjects with a mean pulmonary artery pressure (mPAP) > 25mmHg and a pulmonary artery wedge pressure (PAWP) < 15mmHg at rest, assessed via right heart catheterization.
3. Subjects whose baseline 6-min walk test distance was > 100m and < 450m.

Exclusion Criteria:

1. PAH secondary to any etiology other than those specified in the inclusion criteria.
2. Subjects with congenital heart disease (other than those specified in the inclusion criteria), PAH due to thrombo-embolism, HIV, chronic obstructive airways disease, congestive heart failure.
3. Subjects whose 6-Minute Walk test might have been limited by conditions other than PAH, associated dyspnea or fatigue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Expanded access
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2006-06; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Poland (2):
  - Pfizer Investigational Site, Warsaw
  - Pfizer Investigational Site, Zabrze

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481242&StudyName=To%20Provide%20Sildenafil%20Therapy%20To%20Eligible%20Adult%20Patients%20With%20Pulmonary%20Arterial%20Hypertension%20For%20112%20Weeks

RESULTS

PARTICIPANT FLOW:
Groups:
- Sildenafil 60 mg: Sildenafil 20 mg TID (3 times daily); eligible adult subjects with PAH (pulmonary arterial hypertension)
- Sildenafil 240 mg: Sildenafil 80 mg TID (3 times daily); subjects who completed study A1481142
Period: Overall Study
Arm/Group | Sildenafil 60 mg | Sildenafil 240 mg
Started | 20 | 12
Completed | 12 | 10
Not Completed | 8 | 2
Not completed — Death | 5 | 2
Not completed — Other | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sildenafil 60 mg | Sildenafil 240 mg | Total
Number analyzed (Participants) | 20 | 12 | 32
Age, Customized [Number; unit: participants]
  18 - 44 years | 10 | 6 | 16
  45 - 64 years | 8 | 6 | 14
  >= 65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 26
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Adverse event = any untoward medical occurrence in a subject administered study medication regardless of causality including abnormal test findings, clinically significant signs/symptoms, changes in physical examination findings, hypersensitivity, progression/worsening of underlying disease, and exposure in utero. Serious adverse event = any untoward medical occurrence at any dose that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of hospitalization, or resulted in persistent or significant disability/incapacity or congenital anomaly/birth defect.
Time Frame: Baseline up to 116 Weeks
Population: Safety population: all subjects assumed to have taken at least one dose of study medication. Non-serious adverse events were reported up to 7 days after the last dose of study medication. Serious adverse events were reported up to 28 days after the last dose of study medication.
Measure: Number; unit: participants
Arm/Group | Sildenafil 60 mg | Sildenafil 240 mg
Number analyzed (Participants) | 20 | 12
participants
  AEs | 11 | 8
  SAEs | 8 | 2

ADVERSE EVENTS:
Time Frame: Serious Advserse Events: Baseline up to 28 days after last dose of study medication; Non-serious Adverse Events: Baseline up to 7 days after last dose of study medication
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sildenafil 60 mg | Sildenafil 240 mg
Serious Adverse Events (participants affected / at risk) | 8/20 | 2/12
Other Adverse Events (participants affected / at risk) | 11/20 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil 60 mg (N=20) | Sildenafil 240 mg (N=12)
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 3 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Retinal vein thrombosis (Eye disorders) | 1 | 0
Sudden cardiac death (General disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil 60 mg (N=20) | Sildenafil 240 mg (N=12)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Chest pain (General disorders) | 2 | 1
Fatigue (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 3 | 1
Hepatomegaly (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 2
Neuralgia (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash generalized (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other